CLINICAL TRIAL: NCT04402021
Title: The Effect of Short-term Exercise on Sleep and Daytime Impairment in Adults With Insomnia
Brief Title: Exercise and Insomnia Study: The Effects of 1 Week of Exercise Training on Insomnia Severity
Acronym: Insomni-Ex
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Andrew Kubala, Principle Investigator, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: STUDY20010197
Record Dates: First submitted 2020-05-11; First posted 2020-05-26 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Insomnia Chronic; Insomnia, Primary
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic Exercise (Experimental): Participants randomized to the aerobic exercise group will complete 30 minutes of outdoor walking at a moderate intensity, defined as 50% heart rate reserve from the American College of Sports Medicine (ACSM) exercise prescription recommendations. A 5-minute warm-up and cool-down will occur before and after the 30-minute bout. A Polar H10 heart rate monitor will continuously monitor exercise intensity during the session. Ratings of Perceived Exertion (RPE) will be assessed using the Borg scale (i.e., 6-20 rating system) to indicate perceived exercise effort every 5 minutes during the exercise session. Each session will last approximately 50 minutes.
  Interventions: Behavioral: Outdoor Walking
- Quiet Rest (Other): Participants randomized to this condition will be instructed to watch a nature documentary void of topics related to sleep or exercise. A Polar H10 heart rate monitor will continuously monitor heart rate during the session to mimic the aerobic exercise condition. Participants will not be permitted to complete homework or work during the allotted time to reduce the chance of unintended stimuli. The quiet rest sessions will be 50 minutes in length.
  Interventions: Other: Quiet Rest

INTERVENTIONS:
Behavioral: Outdoor Walking — Unsupervised outdoor walking will be the mode used for moderate-intensity aerobic exercise. The walking intervention will consist of 3 sessions (completed within the span of 7 days) that are conducted in the morning.
  Arms: Aerobic Exercise
Other: Quiet Rest — The quiet rest condition will consist of watching a nature documentary in a quiet room. The quiet rest intervention will consist of 3 sessions (completed within the span of 7 days) that are conducted in the morning.
  Arms: Quiet Rest

SUMMARY:
It has been hypothesized that exercise may have a beneficial effect on sleep quality and insomnia severity in those who have insomnia symptoms as well as those who meet diagnostic criteria for insomnia disorder (e.g., Diagnostic and Statistical Manual 5th edition (DSM-5)). Yet, the studies that have tested this are extremely limited in number and even fewer explore any acute effects of exercise training on subjects who meet diagnostic criteria. Thus, the investigators propose to conduct a randomized parallel design to compare the effects of short-term moderate-intensity aerobic exercise on insomnia severity and measures of sleep in a sample of adults who meet diagnostic criteria for insomnia.

DETAILED DESCRIPTION:
Limited experimental research has explored the effects of acute exercise training (< 1 week of exercise) on sleep and daytime impairment in samples of adults who meet diagnostic criteria for insomnia. In response to the current literature, the investigators aim to better understand the short-term clinical benefit of adopting exercise training in insomnia. Including multiple bouts of exercise in a short time span while measuring sleep with objective and self-reported measures may be more reflective of capturing true acute effects of exercise implementation on insomnia. The investigators propose to conduct a randomized parallel design to compare the effects of short-term moderate-intensity aerobic exercise on insomnia severity and measures of sleep in a sample of adults who meet diagnostic criteria for insomnia. This project will address prior limitations in the area of acute exercise research by utilizing a sample with diagnosed insomnia, assessing multiple nights of sleep, and implementing multiple bouts of exercise stimuli. This project will examine the following aims:

Aim 1: To examine if implementing 1 week of moderate-intensity aerobic exercise improves objective and subjective sleep compared to 1 week without exercise in a sample of adults who meet diagnostic criteria for insomnia.

Aim 2: To examine if implementing 1 week of moderate-intensity aerobic exercise reduces severity of daytime impairment compared to 1 week without exercise in a sample of adults who meet diagnostic criteria for insomnia.

ELIGIBILITY:
Inclusion Criteria:

1. ISI ≥ 10
2. Age 18-55 years
3. Clinically defined Insomnia (i.e., meeting DSM-5 criteria for insomnia disorder)
4. Psychiatric health, aside from treated anxiety and depression determined by participant self-report and instruments described below.

Exclusion Criteria:

1. Unstable acute or chronic medical conditions. Examples include, but are not limited to, central nervous system disorders (e.g., head injury, seizure disorder, multiple sclerosis, tumor), cardiovascular or hemodynamically significant cardiac disease, renal failure, diabetes. Individuals with well-controlled health conditions that do not affect sleep or well-being (e.g., asthma, high blood pressure, diabetes, or ulcers) will not be excluded.
2. Women who are pregnant, nursing, or are planning on becoming pregnant in the next three months.
3. Current untreated major syndromal psychiatric disorders:

   Specific exclusionary self-reports include:
   * Major depressive disorder
   * Dysthymic disorder
   * Bipolar disorder
   * Panic disorder
   * Obsessive compulsive disorder
   * Generalized anxiety disorder
   * Any psychotic disorder
   * Any current substance use disorder

   The investigators will NOT exclude participants for:
   * Untreated subsyndromal symptoms of depression or anxiety and currently treated and stable depression or anxiety disorder.
   * Past episodes of major depressive or anxiety disorder, provided the most recent episode ended at least six months before the diagnostic assessment
   * Simple phobia
   * Social phobia
   * Past eating disorders
   * Past substance use disorders
   * Specific learning disabilities
4. Other current sleep disorders, such as:

   * Insufficient sleep syndrome
   * Circadian rhythm sleep disorders
   * Narcolepsy
   * Restless legs syndrome
   * Obstructive sleep apnea
   * Current night shift work

   Other sleep disorders are diagnosed according to criteria listed in the DSM-5 and the International Classification of Sleep Disorders, 2nd Edition, 2005. These disorders are evaluated using a clinical interview with the Structured Interview for Sleep Disorders.
5. > 0 on the Physical Activity Readiness Questionnaire (PAR-Q+), which represents an inability to safely perform exercise without medical approval or supervision.
6. High risk of sleep-disordered breathing indicated by ≥ 5 'Yes' responses on the STOP-Bang questionnaire, or ≥ 2 + male sex, ≥2 + BMI > 35, or ≥2 + a neck circumference >16 inches (females) or >17 inches (males).
7. Obesity (BMI ≥ 30)
8. Indication of moderate/severe depressive or anxiety symptoms (score ≥ 10 on the Patient Health Questionnaire-9 [PHQ-9] or score ≥ 10 on the 7-item Generalized Anxiety Disorder Questionnaire [GAD-7], respectively)
9. Current treatment for insomnia
10. Suspected circadian rhythm disorder (delayed sleep phase: habitual bedtime ≥ 2:00 am or wake time ≥ 10:00 am; advanced sleep phase: habitual bedtime ≤ 9:00 pm or wake time ≤ 5:00 am)
11. Nocturnal shift-work (i.e., working between 12:00 am and 6:00 am)
12. Physically active (self-report of > 2 sessions/week of structured physical activity or >150 minutes/week of accelerometer-measured bouted moderate to vigorous physical activity)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2020-08-11 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Mean Sleep Efficiency (SE) | Change in SE between baseline and intervention week (approx. 2 weeks)
  Mean SE derived from wrist-worn actigraphy (7 nights of data)
PROMIS Sleep Disturbance Questionnaire (PROMIS SD) score | Change in PROMIS SD between baseline and intervention week (approx. 2 weeks)
  A 5-point Likert scale composed of eight items rated from 1 (not at all, very poor, or never) to 5 (very much, always, or very good) with four items reversed scored. Total raw scores range from 8 to 40 with higher scores indicating greater disturbance. Raw scores will be converted to corresponding T-scores using a published data conversion table.

SECONDARY OUTCOMES:
Insomnia Severity Index (ISI) score | Change in ISI between baseline and intervention week (approx. 2 weeks)
  A 5-point Likert scale is used to rate each item (e.g., 0 = no problem; 4 = very severe problem), yielding a total score ranging from 0 to 28.
PROMIS Sleep Related Impairment Questionnaire (PROMIS SRI) score | Change in PROMIS SRI between baseline and intervention week (approx. 2 weeks)
  A 5-point Likert scale composed of 8 items rated from 1 (not at all) to 5 (very much). One of the eight items (I felt alert when I woke up) is reverse scored. A total score from 8 to 40 is computed with higher scores indicating worse impairment. Total raw scores range from 8 to 40 with higher scores indicating greater disturbance. Raw scores will be converted to corresponding T-scores using a published data conversion table.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Kubala, MS, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual deidentified data that are relevant to the primary aims of the study will be provided to external investigators along with a relevant data dictionary.
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 1 year following peer-reviewed publication of research questions outlined in grant and ending 5 years following publication of study results.
Access Criteria: Data access will be provided to external researchers who provide a methodologically sound proposal for secondary data analysis that is approved by the investigators of the study. Proposals should be directed to the study PI.